CLINICAL TRIAL: NCT05998213
Title: Transfer of Feces in Ulcerative Colitis 2; Improving Efficacy
Brief Title: Transfer of Feces in Ulcerative Colitis 2
Acronym: TURN2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Medical Center Groningen (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Cyriel Y Ponsioen, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL65069.018.18
Record Dates: First submitted 2023-07-12; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Flare; Ulcerative Colitis Acute
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor fecal microbiota transplant (Experimental)
  Interventions: Other: Fecal microbiota transplant
- Autologous fecal microbiota transplant (Placebo Comparator)
  Interventions: Other: Fecal microbiota transplant

INTERVENTIONS:
Other: Fecal microbiota transplant — Frozen FMT via duodenal tube (2 times) and enemas (4 times)
  Other Names: FMT

SUMMARY:
The goal of this placebo-controlled randomised multicenter trial is to evaluate the efficacy and safety of anaerobic prepared donor fecal microbiota transplantation (FMT) compared to autologous FMT in patient with ulcerative colitis.

Participants will receive 4 treatments with frozen FMT via both upper and lower gastro-intestinal route (infusion via duodenal tube and enemas).

Donors are selected based on microbiota profile.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and <70
* Ability to give informed consent
* Established ulcerative colitis with known involvement of the left colon according to the Lennard-Jones criteria
* Partial mayo score of ≥ 3 and calprotectin > 250
* Full Mayo score 5-9
* Endoscopic Mayo score of ≥2 in either the rectum or sigmoid upon screening sigmoidoscopy
* Stable dose of thiopurines or , 5-ASA, or budesonide in preceding 8 weeks.
* Stable dose of budesonide in preceding 2 weeks.
* Prednisone use ≤15mg/day in preceding 2 weeks with a mandatory taper of 5 mg per week starting from week 4.
* Women need to use reliable contraceptives during participation in the study
* Alkaline phosphatase > 1.5 x ULN in the subgroup of PSC/UC patients.

Exclusion Criteria:

* Condition leading to profound immunosuppression

  * For example: HIV, infectious diseases leading to immunosuppression, bone marrow malignancies
  * Use of systemic chemotherapy
  * Child-Pugh B liver cirrhosis
* Anti-TNFα treatment in preceding 2 months
* Vedolizumab treatment in preceding 2 months
* Tofacitinib treatment in preceding 2 months
* Ustekinumab treatment in preceding 2 months
* Cyclosporine treatment in preceding 4 weeks
* Use of Methotrexate in preceding 2 months
* Prednisolone dose > 15 mg/day in preceding 2 weeks
* Use of topical therapy in preceding 2 weeks
* Life expectancy < 12 months
* Difficulty with swallowing
* Use of systemic antibiotics in preceding 4 weeks
* Use of probiotic treatment in preceding 4 weeks
* Positive stool cultures for common enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic e coli)
* Positive C. Difficile stool test
* Positive dual faeces test for pathogenic parasites e.g. Dientamoeba histolytica, Giardia Lamblia, Dientamoeba fragilis, Blastocystis hominis only if microscopically many or very many blastocysts are seen.
* Positive serological test for HIV
* History of surgery:

  * presence of a pouch
  * presence of stoma
* Known intra-abdominal fistula
* Pregnancy or women who give breastfeeding
* Vasopressive medication, icu stay
* Signs of ileus, diminished passage
* Allergy to macrogol or substituents, eg peanuts, shellfish
* Known allergy to iv gadolinium in the subgroup of patients who would be scheduled for MRI liver
* Crohn's disease
* Subject who has any conditions that in the opinion of the investigator, would compromise the safety of the subject or the quality of the data and is an unsuitable candidate for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and endoscopic remission | week 8
  per adapted Mayo: stool frequency subscores (SFS) ≤ 1, rectal bleeding subscore (RBS) =0 and endoscopic subscore ≤ 1.
  The adapted Mayo score has a minimum score of 0 and a maximum score of 9. The 3 subscores (SFS, RBS, and endoscopic subscore) have a minimum of 0 and a maximum score of 3. The adapted Mayo score does not include PGA (physician global assessment), in contrary to the full Mayo score. A higher score reflects worse outcome.

SECONDARY OUTCOMES:
Clinical response | week 8
  Adapted Mayo: decrease from baseline ≥ 2 points and ≥ 30% plus a decrease in RBS ≥ 1 or an absolute RBS ≤ 1.
  The adapted Mayo score has a minimum score of 0 and a maximum score of 9. The 3 subscores (SFS, RBS, and endoscopic subscore) have a minimum of 0 and a maximum score of 3. The adapted Mayo score does not include PGA (physician global assessment), in contrary to the full Mayo score.
Endoscopic response, evaluated by sigmoidoscopy | week 8
  •Proportion of patients with ≥1 point reduction in summed endoscopic Mayo score of both the rectum and sigmoid.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol